CLINICAL TRIAL: NCT04680260
Title: OPTIMIzation of Treatment SElection and Follow up in Oligometastatic Colorectal Cancer - a ctDNA Guided Phase II Randomized Approach
Brief Title: OPTIMIzation of Treatment SElection and Follow up in Oligometastatic Colorectal Cancer
Acronym: OPTIMISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karen-Lise Garm Spindler (Other)
Collaborators: Vejle Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFE2022
Record Dates: First submitted 2020-10-19; First posted 2020-12-22 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: Circulating tumor DNA; Adjuvant chemotherapy; Colorectal cancer; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: An open label 1:1 randomized phase II exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Standard of care (Active Comparator): Standard decision making regarding adjuvant chemotherapy with fluoropyrimidine and oxaliplatin as per institutional standards.
  Interventions: Other: Standard of care
- B: ctDNA guided therapy approach (Experimental): Post ablation ctDNA results will be used for treatment decision.
  Interventions: Other: Circulating tumor DNA guided treatment approach

INTERVENTIONS:
Other: Standard of care — Patients will be offered adjuvant chemotherapy according to standard of care. Follow up will be performed with imaging according to standard guidelines, equal to the experimental arm. Blood samples will be analyzed retrospectively to evaluate the ctDNA status.
  Arms: A: Standard of care
Other: Circulating tumor DNA guided treatment approach — Circulating tumor-marker positivity will lead to escalation with 6 months of intensified chemotherapy consisting of 4 months of FOLFOXIRI followed by 2 months of 5FU monotherapy. Circulating tumor-marker negativity will based on shared decision-making lead to de-escalation i.e. possibilities for observation in patients otherwise eligible for monotherapy or observation/monotherapy in patients, otherwise eligible for combination chemotherapy according to standard of care.
  Arms: B: ctDNA guided therapy approach

SUMMARY:
A study investigating if analysis of circulating tumor DNA (ctDNA) can guide adjuvant treatment in patients with advanced colorectal cancer (CRC)

DETAILED DESCRIPTION:
An open label 1:1 randomized phase II exploratory study investigating use of ctDNA-guided adjuvant chemotherapy compared to standard of care (SOC) after local treatment for metastatic colorectal cancer.

Patients are randomized 1:1 between SOC and ctDNA guided treatment and follow-up.

Escalation therapy comprises standard regimen of Fluorouracil (5-FU), Irinotecan and oxaliplatin (FOLFOXIRI), de-escalation therapy of monotherapy capecitabine or observation only. SOC is per institutional practice, based on national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Radical intended treatment for metastatic spread from CRC, by resection, radiofrequency ablation, stereotactic body radiation therapy (or other experimental local treatment options) not including cytoreductive surgery (CRS) and hyperthermic intra-peritoneal chemotherapy (HIPEC)
* No evidence of further disease based on pre-treatment work-up according to SOC
* Age at least 18 years
* Eastern Cooperative Oncology Group performance status 0-2
* Clinically eligible for adjuvant triple CT at investigators decision.
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy (Absolute neutrophil count ≥1.5x109/l and thrombocytes ≥ 100x109/l. Bilirubin ≤ 1.5 x upper normal value and alanine aminotransferase ≤ 3 x upper normal value, and calculated or measured renal glomerular filtration rate at least 30 mL/min)
* Anticonception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable
* Written and verbally informed consent

Exclusion Criteria:

* Radiological evidence of distant metastasis, by CT- chest, abdomen, and pelvis
* Incapacity, frailty, disability and comorbidity to a degree that according to the investigator is not compatible with triple combination chemotherapy
* Neuropathy National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade > 1
* Other malignant tumor within 5 years except non-melanoma skin cancer or carcinoma in situ cervicis uteri
* Pregnant (positive pregnancy test) or breast feeding women
* Intolerance or allergy to 5FU, leucovorin, oxaliplatin, irinotecan or capecitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Rate | 2 years
  Rate of patients free from recurrent colorectal cancer at 2 years post local treatment

SECONDARY OUTCOMES:
Toxicity of treatment | 6 months post-treatment
  Rate of grade 3-4 toxicity according to CTCAE version 5
Molecular biological response to therapy | 6 months post-treatment
  Rate of patients with lack of detectable tumor DNA in plasma samples
Molecular biological Disease Free Survival | 1 year from inclusion
  Rate of patients with no detectable ctDNA
Time to molecular biological recurrence | 5 years last patient
  Time to molecular biological recurrence is calculated from first time of no detectable DNA until detectable DNA in a samples
Time to radiological recurrence | 5 years last patient
  Time to radiological recurrence is calculated from inclusion until radiological evidence of disease recurrence
Local and distant relapse | 5 years last patient
  Rate of patients with local and distant relapse
Overall survival | 5 years last patient
  Time from inclusion to death from any cause
Quality of life according to EORTC QLQ-CR29 and -C30 | 5 years last patient
  The EORTC QLQ-CR29 is a tumor-specific health related QoL questionnaire module for CRC patients, which complement the EORTC QLQ-C30 questionnaire. Patients indicate their symptoms during the past week(s). Scores can be linearly transformed to a score from 0-100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Quality of life according to EQ-5D-5L | 5 years last patient
  The EQ-5D-5L essentially consists of: the EQ-5D descriptive system and the EQ visual analogue scale. The descriptive system comprises 5 dimensions. Each dimension has 5 levels. The patient is asked to indicate his/her health. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale.
Cost-effectiveness analysis | 5 years last patient
  Economic evaluation of ctDNA guided chemotherapy after curative treatment of metastatic colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, Professor, Principal Investigator — Department of Oncology, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Oncology, Aarhus University Hospital, Aarhus N
  - Department pf Oncology, Vejle Hospital, Vejle